CLINICAL TRIAL: NCT00347750
Title: Pharmacokinetics and Pharmacodynamics of Lopinavir an Anti-HIV Drug in Israeli Ethiopian and Non-Ethiopian Populations
Brief Title: Pharmacokinetics and Pharmacodynamics of an Anti-HIV Drug in Israeli Ethiopian and Non-Ethiopian Populations
Status: Withdrawn | Type: Observational
Why Stopped: lack of participants
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Ministry of Health, Israel (Other Government)
Other Study IDs: 001-2006.CTIL
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2007-04

CONDITIONS: HIV Infection; AIDS
Keywords: Lopinavir; Pharmacokinetic; Pharmacodynamic; Ethiopian population; Caucasian population
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Lopinavir pharmacokinetic/pharmacodynamic analysis

SUMMARY:
The objective of this proposal is based on the assumption that the HIV infected Ethiopian population responded in a different way in comparison to the Caucasian subjects to Lopinavir therapy. Our preliminary data demonstrated that Ethiopian's have different Lopinavir serum concentration in comparison to non-Ethiopian's. For these reasons the plan of this study is to investigate the pharmacokinetic/pharmacodynamic (PK/PD) profile in both populations. The results will allow to establish a better personalised medicine for HIV infected individuals.

DETAILED DESCRIPTION:
The objective of this proposal is based on the assumption that the HIV infected Ethiopian population responded in a different way in comparison to the Caucasian subjects to Lopinavir therapy. Our preliminary data demonstrated that Ethiopian's have different Lopinavir serum concentration in comparison to non-Ethiopian's. For these reasons the plan of this study is to investigate the pharmacokinetic/pharmacodynamic (PK/PD) profile in both populations. The results will allow to establish a better personalised medicine for HIV infected individuals.

ELIGIBILITY:
Inclusion Criteria:

* All HIV infected Ethiopian and Non-Ethiopian subjects
* AIDS diseased Ethiopian and Non-Ethiopian individuals

Exclusion Criteria:

* Individuals who are unable to sign the informed concent
* Individuals unable to take oral medications
* Individuals who described Lopinavir allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Krivoy, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel